CLINICAL TRIAL: NCT06250543
Title: Evaluation of Intradetrusor AbobotulinumtoxinA and IncobotulinumtoxinA Efficacy and Safety in Women With Overactive Bladder and Urge Urinary Incontinence and the Value of Local Anesthesia for Pain Reduction
Brief Title: Evaluation of Intradetrusor AbobotulinumtoxinA and IncobotulinumtoxinA in Women With Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Niko Kavcic (Other)
Responsible Party: Sponsor-Investigator, Niko Kavcic, MD, University Medical Centre Maribor
Organization: University Medical Centre Maribor (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRP-2018-01-14
Record Dates: First submitted 2024-01-18; First posted 2024-02-09 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Overactive Bladder
Keywords: botulinum toxin; overactive bladder; abobotulinumtoxinA; incobotulinumtoxinA; local anesthesia
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Patients were randomized to receive 20 intradetrusor injections of either 300 U AbobotulinumtoxinA or 100 U IncobotulinumtoxinA. They were further randomized to receive either local anesthesia (40 ml of 1% lidocaine solution) or placebo before botulinum toxin injection.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AbobotulinumtoxinA and lidocaine (Other): The bladder was instilled with 40 ml of 1% lidocaine solution using a 16Fr urethral Foley catheter.
  30 minutes afterwards patients received 300 units of AbobotulinumtoxinA using rigid cystoscopy. Normal saline was used to dilute the vial to 20 ml. A total of 20 evenly distributed intradetrusor injections, 1 ml per site, were performed, 2 of them included the trigone area.
  Interventions: Drug: AbobotulinumtoxinA 300 UNT; Drug: Lidocain
- AbobotulinumtoxinA and placebo (Other): The bladder was instilled with 40 ml of 0.9% NaCl solution using a 16Fr urethral Foley catheter.
  30 minutes afterwards patients received 300 units of AbobotulinumtoxinA using rigid cystoscopy. Normal saline was used to dilute the vial to 20 ml. A total of 20 evenly distributed intradetrusor injections, 1 ml per site, were performed, 2 of them included the trigone area.
  Interventions: Drug: AbobotulinumtoxinA 300 UNT; Other: placebo
- IncobotulinumtoxinA and lidocaine (Other): The bladder was instilled with 40 ml of 1% lidocaine solution using a 16Fr urethral Foley catheter.
  30 minutes afterwards patients received 100 units of IncobotulinumtoxinA using rigid cystoscopy. Normal saline was used to dilute the vial to 20 ml. A total of 20 evenly distributed intradetrusor injections, 1 ml per site, were performed, 2 of them included the trigone area.
  Interventions: Drug: IncobotulinumtoxinA 100 UNT; Drug: Lidocain
- IncobotulinumtoxinA and placebo (Other): The bladder was instilled with 40 ml of 0.9% NaCl solution using a 16Fr urethral Foley catheter.
  30 minutes afterwards patients received 100 units of IncobotulinumtoxinA. using rigid cystoscopy. Normal saline was used to dilute the vial to 20 ml. A total of 20 evenly distributed intradetrusor injections, 1 ml per site, were performed, 2 of them included the trigone area.
  Interventions: Drug: IncobotulinumtoxinA 100 UNT; Other: placebo

INTERVENTIONS:
Drug: AbobotulinumtoxinA 300 UNT — 20 evenly distributed intradetrusor injections, 1 ml per site, were performed
  Arms: AbobotulinumtoxinA and lidocaine; AbobotulinumtoxinA and placebo
Drug: IncobotulinumtoxinA 100 UNT — 20 evenly distributed intradetrusor injections, 1 ml per site, were performed
  Arms: IncobotulinumtoxinA and lidocaine; IncobotulinumtoxinA and placebo
Drug: Lidocain — 30 minutes before the procedure the bladder was instilled with 40 ml of 1% lidocaine solution using a 16Fr urethral Foley catheter
  Arms: AbobotulinumtoxinA and lidocaine; IncobotulinumtoxinA and lidocaine
Other: placebo — 30 minutes before the procedure the bladder was instilled with 40 ml of 0.9% NaCl solution
  Arms: AbobotulinumtoxinA and placebo; IncobotulinumtoxinA and placebo

SUMMARY:
A randomized, single blind, non-inferiority clinical study was performed evaluating the efficacy and safety of AbobotulinumtoxinA vs. IncobotulinumtoxinA intradetrusor injections in women with overactive bladder and urge urinary incontinence. Also the effect of local anesthesia on pain level of the procedure was assessed.

DETAILED DESCRIPTION:
In the described prospective, clinical trial, approved by the National Medical Ethics Committee (protocol number: 0120-44/2018/5; date of approval: 22/02/2018), female patients were enrolled, followed by signed informed consent.

Before treatment patients underwent history and physical examination. Before botulinum toxin injection each patient completed three questionnaires, UDI-6 (Urogenital Distress Inventory), IIQ-7 (Incontinence Impact Questionnaire), I-QOL (Incontinence Quality of Life). The total score of each questionnaire was considered. Before botulinum toxin injection, urinalysis was performed to check for a urinary tract infection (UTI). For those presenting with UTI, treatment was postponed until the UTI was treated and a repeat urinalysis was performed. Nitrofurantoin 100 mg twice daily per os was given prophylactically on the day of the procedure. Patients were randomised to receive either 300 units of AbobotulinumtoxinA (Dysport®) or 100 units of IncobotulinumtoxinA (Xeomin®). They were further randomised to receive local anesthesia or placebo. 30 minutes before the procedure the bladder was instilled with either 40 ml 1% lidocaine solution using a 16Fr urethral Foley catheter or with 40 ml 0.9% NaCl solution. All patients received urethral lubrication gel. Using rigid cystoscopy, normal saline was used to dilute the vial to 20 ml. A total of 20 evenly distributed intradetrusor injections, 1 ml per site, were performed, 2 of them included the trigone area. During the procedure the patients graded the pain level of every injection on a Visual Analog Scale (VAS). All patients were treated in an outpatient clinic and by one experienced surgeon.

After 1 to 2 weeks patients were seen for evaluation of systemic side effects, physical examination, measurement of residual urine and urinalysis to eventually diagnose and treat a urinary tract infection. After 4 months patients were seen to evaluate the treatment result and complete the questionnaires, IIQ-7, UDI-6, patient satisfaction survey and I-QOL. Side effects were monitored for 5 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* female, age between 18 and 90, presence of urinary urgency with urgency urinary incontinence, residual urine below 150 ml, previous non-pharmacological conservative treatments (e.g., pelvic floor muscle training) inefficiency, anticholinergic or beta-3 agonist treatment inefficiency.

Exclusion Criteria:

* patients that already have received treatment with botulinum toxin, pregnancy or breast- feeding and any diseases or functional abnormalities that might affect bladder function. Patients with stress urinary incontinence.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of Intradetrusor AbobotulinumtoxinA and IncobotulinumtoxinA | 5 months
  Questionnaire scores of UDI-6 (Urogenital Distress Inventory), IIQ-7 (Incontinence Impact Questionnaire) and I-QOL (Incontinence Quality of Life) will be evaluated before and after the procedure for non-inferiority of the two drugs.

SECONDARY OUTCOMES:
The Value of Local Anesthesia for Pain Reduction | The day of procedure
  During the procedure the patients graded the pain level of every injection on a Visual Analog Scale (VAS). The total score of each questionnaire will be evaluated for non-inferiority of placebo in comparison to local anesthesia.
Safety of Intradetrusor AbobotulinumtoxinA and IncobotulinumtoxinA | 5 months
  Frequency of adverse events (urinary retention, urinary tract infection)

CONTACTS AND LOCATIONS:
Overall Officials: Niko Kavčič, MD, Principal Investigator — University Medical Centre Maribor
Locations (1):
- University Medical Centre Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
We intend to publish a research article in 2024. All supporting information will be shared with the journal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We intend to publish a research article in 2024. All supporting information will be shared with the journal.
Access Criteria: Access will be provided by the journal.

REFERENCES:
- [Background] Giannantoni A, Gubbiotti M, Rubilotta E, Balzarro M, Antonelli A, Bini V. IncobotulinumtoxinA versus onabotulinumtoxinA intradetrusor injections in patients with neurogenic detrusor overactivity incontinence: a double-blind, randomized, non-inferiority trial. Minerva Urol Nephrol. 2022 Oct;74(5):625-635. doi: 10.23736/S2724-6051.21.04227-2. Epub 2021 Mar 26. PMID 33769020
- [Background] Lange S, Koch M, Lange R, Husslein H, Umek W, Bodner-Adler B. Perioperative Techniques for the Use of Botulinum Toxin in Overactive Bladder: Results of a Multinational Online Survey of Urogynecologists in Germany, Austria, and Switzerland. J Clin Med. 2023 Feb 12;12(4):1462. doi: 10.3390/jcm12041462. PMID 36835999